CLINICAL TRIAL: NCT01298596
Title: Impact of Cryotherapy Versus Loop Electrosurgical Excision Procedure (LEEP) on Recurrence of Cervical Intraepithelial Neoplasia and HIV-1 Cervical Shedding Among HIV-positive Women
Brief Title: Cryotherapy vs. LEEP to Treat Cervical Intraepithelial Neoplasia (CIN) 2/3 Among HIV-positive Women
Acronym: PHE-LEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Nairobi (Other); International Agency for Research on Cancer (Other)
Responsible Party: Principal Investigator, Michael Chung, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35995-J; KE.09.0238 (Other: Kenya Ethical Review Committee)
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryotherapy (Experimental): Cryotherapy procedure involves using a cryoprobe and carbon dioxide or nitrous oxide gas to freeze the diseased part of the cervix
  Interventions: Procedure: Cryotherapy
- Loop Electrosurgical Excision Procedure (Experimental): Loop Electrosurgical Excision Procedure (LEEP) uses a low-voltage electrified wire loop to cut out diseased part of cervix
  Interventions: Procedure: Loop Electrosurgical Excision Procedure (LEEP)

INTERVENTIONS:
Procedure: Loop Electrosurgical Excision Procedure (LEEP) — LEEP procedure uses a low-voltage electrified wire loop to cut out diseased part of cervix
  Other Names: LEEP
  Arms: Loop Electrosurgical Excision Procedure
Procedure: Cryotherapy — Cryotherapy procedure involves using a cryoprobe and carbon dioxide or nitrous oxide gas to freeze the diseased part of the cervix
  Arms: Cryotherapy

SUMMARY:
The purpose of this study is to compare the rate of recurrence of cervical intraepithelial neoplasia among HIV-positive women receiving cryotherapy versus LEEP over 2 years of follow-up and to compare the shedding of HIV-1 from the cervix between HIV-positive women receiving cryotherapy versus LEEP over 3 weeks of follow-up.

DETAILED DESCRIPTION:
The recent scale-up of antiretroviral treatment programs in resource-limited settings provides an unprecedented opportunity to implement a comprehensive cervical cancer screening and treatment program for women who, by virtue of having HIV, are at significant risk for cervical disease. Unfortunately, even if screening is offered free of charge to millions of women living with HIV, it is unclear which treatment modality for pre-cancerous cervical lesions will be most effective since HIV appears to affect outcomes of treatment by increasing the recurrence and severity of cervical disease. Cervical treatment may also increase shedding of HIV from the cervix which may put discordant couples at risk and possibly spread HIV more widely. This study proposes to randomize HIV-positive women with cervical intraepithelial neoplasia grade 2 and 3 (CIN 2 and 3) to cryotherapy vs. loop electrosurgical excision procedure (LEEP) and measure the recurrence of cervical disease in each group over 2-years of follow-up as well as HIV shedding from the cervix for 6 weeks after treatment.

Our hypothesis is that compared to cryotherapy, LEEP is significantly more likely to prevent recurrence of cervical lesions over 2 years of follow-up and less likely to cause shedding of HIV-1 from the cervix over 3 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive receiving care at the Coptic Hope Center
* Not pregnant by clinical examination or history
* Have an intact cervix
* Have not received prior cervical treatment
* Do not have a history of a bleeding disorder
* Are above 18 years of age

Exclusion Criteria:

* HIV-negative
* Male
* Below 18 years of age
* Pregnant by clinical examination or history
* Post-hysterectomy
* Post-cervical cancer treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chung, MD, Principal Investigator — University of Washington
Locations (1):
- Coptic Hospital, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung MH, De Vuyst H, Greene SA, Mugo NR, Querec TD, Nyongesa-Malava E, Cagle A, Sakr SR, Luchters S, Temmerman M, Unger ER, McGrath CJ. Human Papillomavirus Persistence and Association With Recurrent Cervical Intraepithelial Neoplasia After Cryotherapy vs Loop Electrosurgical Excision Procedure Among HIV-Positive Women: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2021 Oct 1;7(10):1514-1520. doi: 10.1001/jamaoncol.2021.2683. PMID 34351377
- [Derived] Greene SA, De Vuyst H, John-Stewart GC, Richardson BA, McGrath CJ, Marson KG, Trinh TT, Yatich N, Kiptinness C, Cagle A, Nyongesa-Malava E, Sakr SR, Mugo NR, Chung MH. Effect of Cryotherapy vs Loop Electrosurgical Excision Procedure on Cervical Disease Recurrence Among Women With HIV and High-Grade Cervical Lesions in Kenya: A Randomized Clinical Trial. JAMA. 2019 Oct 22;322(16):1570-1579. doi: 10.1001/jama.2019.14969. PMID 31638680
- [Derived] Greene SA, McGrath CJ, Lehman DA, Marson KG, Trinh TT, Yatich N, Nyongesa-Malava E, Kiptinness C, Richardson BA, John-Stewart GC, De Vuyst H, Sakr SR, Mugo NR, Chung MH. Increased Cervical Human Immunodeficiency Virus (HIV) RNA Shedding Among HIV-Infected Women Randomized to Loop Electrosurgical Excision Procedure Compared to Cryotherapy for Cervical Intraepithelial Neoplasia 2/3. Clin Infect Dis. 2018 May 17;66(11):1778-1784. doi: 10.1093/cid/cix1096. PMID 29272368

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cryotherapy | Loop Electrosurgical Excision Procedure
Started | 200 | 200
Completed | 172 | 167
Not Completed | 28 | 33
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 5 | 3
Not completed — Lost to Follow-up | 6 | 14
Not completed — Referred for further management | 16 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryotherapy | Loop Electrosurgical Excision Procedure | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Categorical [Count of Participants; unit: Participants] — Population: Not all women provided age or a date of birth at baseline
  Participants
    number analyzed (Participants) | 194 | 189 | 383
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 194 | 189 | 383
    >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Not all women provided age or a date of birth at baseline
  years
    number analyzed (Participants) | 194 | 189 | 383
    (all) | 38.2 [32.0 to 42.5] | 37.4 [31.7 to 44.9] | 37.4 [31.7 to 43.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 200 | 400
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 200 | 200 | 400
Previously screened for cervical cancer [Count of Participants; unit: Participants] — Population: Some women were uncertain of prior screening status
  Participants
    number analyzed (Participants) | 189 | 189 | 378
    (all) | 65 | 55 | 120

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of Cervical Intraepithelial Neoplasia Among HIV-positive Women
Description: Rate of recurrence of cervical intraepithelial neoplasia among HIV-positive women receiving cryotherapy versus LEEP over 2 years of follow-up
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cryotherapy | Loop Electrosurgical Excision Procedure
Number analyzed (Participants) | 200 | 200
Participants | 60 | 37

2. Secondary Outcome: Shedding of HIV-1 From the Cervix Between HIV-positive Women
Description: Shedding of HIV-1 from the cervix between HIV-positive women receiving cryotherapy versus LEEP between baseline and weeks 1, 2, and 3 of follow-up
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: change in log10 cps HIV RNA per swab
Arm/Group | Cryotherapy | Loop Electrosurgical Excision Procedure
Number analyzed (Participants) | 200 | 200
change in log10 cps HIV RNA per swab
  Baseline and Week 1 | -0.02 [-0.11 to 0.06] | 0.10 [0.02 to 0.18]
  Baseline and Week 2 | 0.07 [-0.02 to 0.16] | 0.25 [0.14 to 0.37]
  Baseline and Week 3 | 0.05 [-0.05 to 0.14] | 0.26 [0.14 to 0.38]

ADVERSE EVENTS:
Time Frame: 24 months
Description: We used Division of AIDS Table for Grading the Severity of Adult Adverse Events version 1.0.
  Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
Arm/Group | Cryotherapy | Loop Electrosurgical Excision Procedure
Serious Adverse Events (participants affected / at risk) | 5/200 | 2/200
Other Adverse Events (participants affected / at risk) | 2/200 | 0/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryotherapy (N=200) | Loop Electrosurgical Excision Procedure (N=200)
HIV complications (Infections and infestations) | 5 (5) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryotherapy (N=200) | Loop Electrosurgical Excision Procedure (N=200)
Related to procedure (Surgical and medical procedures) | 2 (2) | 0 (0) — post-operative bleeding

LIMITATIONS AND CAVEATS:
1) Conducted in a single center with one clinician administering all procedures 2) Human papillomavirus-type specific results not available 3) HIV factors vary with time 4) Longer follow-up is necessary 5) Imbalance in cervical HIV RNA at baseline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT01298596/Prot_SAP_ICF_000.pdf